CLINICAL TRIAL: NCT04206722
Title: Efficiency of Shock-wave Therapy in Symptomatic Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ciubean Alina Deniza, Principal investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversitateaMFHIL
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Extracorporeal Shockwave Therapy; Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Shock Wave therapy on the affected hip, for 10 days, 1 application every 2 days
  Interventions: Device: Shock Wave Therapy
- Control group (Active Comparator): Ultrasound therapy on the affected hip, for 10 days, 1 application daily
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Shock Wave Therapy — Shock Wave therapy - hip osteoarthritis program
  Arms: Treatment group
Device: Ultrasound — Ultrasound 0.7W/cm2
  Arms: Control group

SUMMARY:
The objectives of treatment in hip osteoarthritis are pain relief, improve joint range of motion and muscle force, gait rehabilitation, patient education and socio-professional reintegration.The non-pharmacological and non-surgical methods include certain types of physical therapy: massage, heat, ultrasound, laser, shockwave therapy. Few studies have been conducted so far for outcome measurement in symptomatic hip osteoarthritis.

DETAILED DESCRIPTION:
The objectives of treatment in hip osteoarthritis are pain relief, improve joint range of motion and muscle force, gait rehabilitation, patient education and socio-professional reintegration.The non-pharmacological and non-surgical methods include certain types of physical therapy: massage, heat, ultrasound, laser, shockwave therapy. Among them, shockwave therapy is not a new treatment method, and seems to be effective in rotator cuff pathology, tennis elbow, and also on knee osteoarthritis, but few studies have been conducted so far for outcome measurement in symptomatic hip osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral hip osteoarthritis

Exclusion Criteria:

* other disorders that are contraindications for shockwave or ultrasound application

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change from baseline Visual Analogue Scale (VAS) score at 10 days and 30 days | at baseline, after 10 days, after 30 days
  10mm to 100mm, higher scores mean a worse outcome

SECONDARY OUTCOMES:
change from baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score at 10 days and 30 days | at baseline, after 10 days, after 30 days
  24-item questionnaire for osteoarthritis, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Irsay Laszlo, MD, PhD, Study Director — University of Medicine and Pharmacy Iuliu Hatieganu

IPD SHARING:
Plan to Share IPD: Undecided
upon request